CLINICAL TRIAL: NCT00493324
Title: An Open-Label Phase 4 Study in Adult Patients With Chronic Plaque Psoriasis to Evaluate the Immune Response to Pneumococcal Vaccine in Subjects Treated With Alefacept
Brief Title: Study to Evaluate the Immune Response to Pneumococcal Vaccine in Alefacept-treated Adults With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0485-CL-0003
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: psoriasis; alefacept; polyvalent pneumococcal vaccine; Immunization
MeSH Terms: conditions — Psoriasis | interventions — Alefacept; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: alefacept; Drug: polyvalent pneumococcal vaccine

INTERVENTIONS:
Drug: alefacept — Intramuscular
  Other Names: Amevive®; ASP0485
Drug: polyvalent pneumococcal vaccine — Injection
  Other Names: PNEUMOVAX® 23

SUMMARY:
A vaccine causes the immune system to produce antibodies (immune response) to specific germs to protect the patient. This study evaluates the immune response to the pneumococcal vaccine in adults with Alefacept-treated chronic plaque psoriasis.

DETAILED DESCRIPTION:
This is a 1 arm study designed to evaluate the immune response to pneumococcal vaccine in adults with Alefacept-treated chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has chronic plaque psoriasis
* Subject has at least 5% body surface area affected with psoriasis

Exclusion Criteria:

* Skin disorder other than plaque psoriasis in affected area
* Previously immunized with any pneumococcal vaccine
* Subject has pustular or erythrodermic psoriasis
* Subject is immunocompromised
* Six or more herpes simplex virus outbreaks per year
* History or malignancy, chronic serious infection or hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects with at least a 2-fold increase in 2 or more of 5 pneumococcal antibody titers. | 12 weeks

SECONDARY OUTCOMES:
The number and percentage of subjects with an antibody response to pneumococcal antigens | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (6):
- United States (4):
  - Birmingham, Alabama
  - San Diego, California
  - New York, New York
  - Cleveland, Ohio
- Canada (2):
  - St. John's, Newfoundland and Labrador
  - Markham, Ontario

REFERENCES:
- [Background] Lynde C, Krell J, Korman N, Mathes B; Vaccine Study Investigators. Immune response to pneumococcal polysaccharide vaccine in adults with chronic plaque psoriasis treated with alefacept. J Am Acad Dermatol. 2011 Oct;65(4):799-806. doi: 10.1016/j.jaad.2010.04.040. Epub 2011 Mar 30. PMID 21453987